CLINICAL TRIAL: NCT04196361
Title: Ultrasonography for Prediction of Extubation Success: a Holistic Approach
Acronym: APEX
Status: Completed | Type: Observational
Sponsor: Amsterdam UMC, location VUmc (Other)
Responsible Party: Principal Investigator, Jasper M Smit, MD, Medical Doctor, Amsterdam UMC, location VUmc
Other Study IDs: 2016.465
Record Dates: First submitted 2019-12-09; First posted 2019-12-12 (Actual); Last update posted 2019-12-12 (Actual); Status verified 2019-12

CONDITIONS: Exutbation Failure; Mechanical Ventilation
Keywords: Ultrasound; Diaphragm; Holistic; Extubation
MeSH Terms: interventions — Ultrasonography

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Ventilated72h: Patient that were ventilated for at least 72 hours
  Interventions: Diagnostic Test: Ultrasound

INTERVENTIONS:
Diagnostic Test: Ultrasound — Point of care ultrasound as part of routine physical examination

SUMMARY:
This study evaluates thickening fraction alone and together with other ultrasound parameters of heart and lungs as predictors for extubation outcome

DETAILED DESCRIPTION:
Weaning patients in the intensive care unit (ICU) from the mechanical ventilator is a critical period and accounts for 40% of the duration of mechanical ventilation itself. Weaning failure includes failing the initial spontaneous breathing trial (SBT) and patients with extubation failure. Extubation failure is defined as reintubation or need for rescue non-invasive ventilation within 48 hours following extubation. Patients failing extubation experience increased time spent on the mechanical ventilator and even increased mortality rates. Given these risks, predicting readiness for extubation is of key importance in the ICU.

Studies have shown, that US is a viable tool for routine use due to its bedside availability and non-invasiveness, while still maintaining excellent predictive values for its respective applications. For this reason, over the past years, critical care ultrasonography (US) has become an important part of routine bedside assessment Lately, the diaphragm has been studied extensively, due to its strong role in sustaining spontaneous breathing. Especially predicting extubation outcomes

has become a great field of interest and different studies have been conducted on this topic. Currently, indices such as diaphragm thickening (Tdi), diaphragm thickness (Tdi%) and diaphragm motion are the most frequently used parameters. Of these, thickening fraction seems to be the most promising to predict successful extubation.

However, all of the studies conducted, solely looked at diaphragm function and compared them to current standards such as the rapid shallow breathing index, while disregarding other factors strongly correlated to extubation failure, e.g. respiratory and cardiac function, as proposed by Mayo et al. Taking heart and lung function into account as well seems to be an interesting approach, because additional measurements could possibly improve predictive value while putting no further burden on the patient. Furthermore, both heart and lungs can be assessed quickly and easily by ultrasound. Cardiac parameters that are potentially useful are left ventricular function, mitral diastolic inflow and cardiac output. Regarding the lungs, pleural effusion is associated with rate of success for extubation. Effusion is detected easily and recent studies have shown, that in an ICU setting a simple 8 region protocol is sufficient to detect extra vascular lung water.

The investigators hypothesise that a holistic US approach, including measurements of heart, lungs and diaphragm, will be superior to the core diagnostic parameters of the diaphragm in predicting extubation success in mechanically ventilated critical care patients.

ELIGIBILITY:
Inclusion Criteria:

* Ventilated for > 72 hours
* Passed spontaneous breathing trial

Exclusion Criteria:

* Planned NIV
* Palliative Extubation
* Tracheostomy
* Paraplegia above Th 8

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population consisted of adult (>18 years) patients, admitted to the ICU and ventilated for at least 72h.
Sampling Method: Probability Sample
Enrollment: 83 (Actual)
Dates: Start 2016-09-01 (Actual); Primary Completion 2019-11-29 (Actual); Study Completion 2019-12-02 (Actual)

PRIMARY OUTCOMES:
Sensitivity | 48 hours
  Sensitivity of thickening fraction for extubation failure
Specificity | 48 hours
  Specificity of thickening fraction for extubation failure
Area under the Curve | 48 hours
  Area under the receiver operator curve
Correlation of ultrasound variables with extubation outcome | 48 hours
  Correlation of ultrasound variables with extubation outcome through (logistic)regression analysis.

IPD SHARING:
Plan to Share IPD: Yes
Upon we request we can share our data to assist other researchers with interest in this field of research.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: After publication in a peer reviewed journal

REFERENCES:
- [Derived] Haaksma ME, Smit JM, Heldeweg M, Nooitgedacht JS, Atmowihardjo LN, Jonkman AH, de Vries HJ, Lim EH, Steenvoorden T, Lust E, Girbes AR, Heunks LM, Tuinman PR. Holistic Ultrasound to Predict Extubation Failure in Clinical Practice. Respir Care. 2021 Jun;66(6):994-1003. doi: 10.4187/respcare.08679. Epub 2021 Apr 13. PMID 33850048